CLINICAL TRIAL: NCT01296971
Title: Open-label, Multicenter, Non-Comparative Prospective Study to Assess the Safety of Individualized Combination Therapy With Ribavirin And Peginterferon Alfa-2a (40 kD) in Patients With Chronic Hepatitis C (CHC) (MASTER Study)
Brief Title: A Study of the Safety of Individualized Combination Therapy With Copegus (Ribavirin) and Pegasys (Peginterferon Alfa-2a) in Patients With Chronic Hepatitis C (MASTER)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: study was not started due to an administrative reason on the part of the local Health Authority
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML25246
Record Dates: First submitted 2010-12-21; First posted 2011-02-16 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

ARMS (3):
- A (Experimental): genotype 1, treatment-naive
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin [Copegus]
- B (Experimental): genotype 2 and 3, treatment-naive
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin [Copegus]
- C (Experimental): all genotypes, non-responders or relapses
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin [Copegus]

INTERVENTIONS:
Drug: peginterferon alfa-2a [Pegasys] — 180 mcg sc weekly
Drug: ribavirin [Copegus] — 1'000/1'200 mg daily orally, 24 - 72 weeks
  Arms: A; C
Drug: ribavirin [Copegus] — 800 mg daily orally, 16 - 48 weeks
  Arms: B

SUMMARY:
This open-label, non-comparative study will assess the safety and tolerability of individualized combination therapy with Copegus (ribavirin) and Pegasys (peginterferon alfa-2a) in patients with chronic hepatitis C. Patients with hepatitis C virus (HCV) genotype 1 (Group A) will receive Copegus 1'000 mg or 1'200 mg daily orally for 24-72 weeks. For patients with genotype 2 or 3 HCV (Group B) the Copegus dose will be 800 mg daily for 16-48 weeks. Patients who had previously received standard or pegylated interferons but were non-responders or with relapse (Group C) will receive Copegus 1'000 mg or 1'200 mg daily for up to 72 weeks. Concomitant therapy with Pegasys 180 mcg subcutaneously weekly will be given to all patients. Anticipated time on study treatment is up to 72 weeks with a 24-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Chronic hepatitis C
* Measurable serum HVC RNA levels
* Compensated liver disease (Child-Pugh class A)
* Treatment-naive for standard or pegylated interferons, or non-responder or relapsing

Exclusion Criteria:

* Concomitant hepatitis A or B
* History of chronic liver disease not caused by hepatitis C virus
* Hepatocellular carcinoma
* History or signs of esophageal varices haemorrhage or other conditions indicative of decompensated liver disease
* Treatment with any systemic anti-tumor or immunomodulatory agent (including steroids at doses exceeding physiological ones, and radiotherapy) within 6 months prior to first dose of study drug
* Pregnant or lactating women, or men whose partners are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Safety of individualized Copegus treatment in combination with Pegasys: Adverse events | up to 96 weeks
Influence of dose reductions in case of adverse events on sustained virological response (HCV-RNA) | up to 96 weeks

SECONDARY OUTCOMES:
Virological response/sustained virological response (serum HCV RNA levels) | 24 weeks after treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche